CLINICAL TRIAL: NCT07079930
Title: Safety and Psychological Effects of Psilocybin and D-Serine Formulation in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Ps-PD-24-01-HMO-CTIL
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers
Keywords: psilocybin D-Serine healthy volunteers
MeSH Terms: interventions — Psilocybin; Physical Examination; Vital Signs; Blood Cell Count; Urinalysis; Electroencephalography; Psychiatric Status Rating Scales

STUDY DESIGN:
Intervention Model Description: The study will include 2 cohorts:
  First cohort of 5 participants will be recruited and administered a single dose of 15 mg of Psilocybin and 5 gr of D-Serine. Safety data will be collected, and an interim safety report will be submitted to the Ethics Committee (EC).
  Following administration to the initial cohort, safety and tolerability will be evaluated, and if no significant concerns are identified, the second cohort will be enrolled to receive a higher dose in order to determine the optimal dosage
  The second cohort of 5 participants will receive an increased one time dose of 25 mg of Psilocybin and 7 gr of D-Serine to determine the effective dose.
  The following visits will be conducted for both cohorts: Screening, Preparation, Administration (Day 1), and follow-up visits on Day 2, Day 7, Day 28, and Day 84.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 15 mg of Psilocybin and 5 gr of D-Serine (Experimental): The investigational drug, 15 mg of Psilocybin and 5 g of D-Serine, will be administered as a single oral dose in solution form.
  Interventions: Drug: Psilocybin and D-Serine; Diagnostic Test: Physical Examination; Diagnostic Test: Vital signs; Diagnostic Test: ECG test; Diagnostic Test: Comprehensive Blood Panel; Diagnostic Test: Complete Blood Count; Diagnostic Test: Urinalysis; Diagnostic Test: Urine Toxicology Screen; Diagnostic Test: A pregnancy Urine test; Diagnostic Test: Electroencephalogram; Diagnostic Test: Plasma Amino Acid Levels; Diagnostic Test: Plasma Inflammation Markers; Diagnostic Test: Plasma Brain-Derived Neurotrophic Facto; Other: Mini International Neuropsychiatric Interview; Other: Family Psychiatric History Assessment; Other: Beck Depression Inventory; Other: State-Trait Anxiety Inventory; Behavioral: Profile of Mood States; Behavioral: Subjective Units of Distress Scale; Other: Five-Dimensional Altered States of Consciousness questionnaire; Behavioral: Integration
- 25 mg of Psilocybin and 7 gr of D-Serine (Experimental): The investigational drug, 25 mg of Psilocybin and 7 g of D-Serine, will be administered as a single oral dose in solution form.
  Interventions: Drug: Psilocybin and D-Serine; Diagnostic Test: Physical Examination; Diagnostic Test: Vital signs; Diagnostic Test: ECG test; Diagnostic Test: Comprehensive Blood Panel; Diagnostic Test: Complete Blood Count; Diagnostic Test: Urinalysis; Diagnostic Test: Urine Toxicology Screen; Diagnostic Test: A pregnancy Urine test; Diagnostic Test: Electroencephalogram; Diagnostic Test: Plasma Amino Acid Levels; Diagnostic Test: Plasma Inflammation Markers; Diagnostic Test: Plasma Brain-Derived Neurotrophic Facto; Other: Mini International Neuropsychiatric Interview; Other: Family Psychiatric History Assessment; Other: Beck Depression Inventory; Other: State-Trait Anxiety Inventory; Behavioral: Profile of Mood States; Behavioral: Subjective Units of Distress Scale; Other: Five-Dimensional Altered States of Consciousness questionnaire; Behavioral: Integration

INTERVENTIONS:
Drug: Psilocybin and D-Serine — A single administration of the drug, with dosage divided as follows:
  Cohort 1: 15 mg of Psilocybin and 5 gr of D-Serine Cohort 2: 25 mg of Psilocybin and 7 gr of D-Serine
Diagnostic Test: Physical Examination — The physical examination will include diagnosis and documentation of any significant clinical abnormalities or diseases. It will be performed during the baseline rating visit (preparation phase).
Diagnostic Test: Vital signs — Vital sign measurements (blood pressure, pulse, and oxygen saturation) will be taken at screening, preparation, baseline rating, administration day, day 2, day 28, and day 84.
  Vital signs will be assessed at the following time points on the administration day and on day 2: pre-administration, and at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 20, and 24 hours post-administration.
Diagnostic Test: ECG test — A 12-lead ECG will be performed to rule out underlying cardiac abnormalities. An ECG will be conducted for each patient during the screening and Day 2 visits.
Diagnostic Test: Comprehensive Blood Panel — A comprehensive blood panel will be performed to assess kidney and liver function, electrolyte balance, and glucose levels.
  It will be conducted during the Screening visit, and on Day 2, Day 28, and Day 84.
  Other Names: SMAC-20
Diagnostic Test: Complete Blood Count — Complete Blood Count will be performed to check for hematological abnormalities.
  It will be conducted during the Screening visit, and on Day 2, Day 28, and Day 84.
  Other Names: CBC
Diagnostic Test: Urinalysis — Urinalysis will be conducted during the Screening visit, and on Day 2, Day 28, and Day 84.
Diagnostic Test: Urine Toxicology Screen — Urine Toxicology Screen will be performed to rule out illicit drug use. It will be conducted during the Screening visit, and on Day 2, Day 28, and Day 84.
Diagnostic Test: A pregnancy Urine test — A urine pregnancy test will be performed for women of childbearing potential only. It will be conducted during the screening and baseline rating visits. If the urine test is positive, a serum β-hCG test will be performed for confirmation.
Diagnostic Test: Electroencephalogram — EEG will be performed during the baseline rating scale and Day 7 visits to evaluate brain activity
  Other Names: EEG
Diagnostic Test: Plasma Amino Acid Levels — The following blood test parameters - D-Serine, L-Serine, and Glycine - will be assessed during the Screening and Day 28 visits.
Diagnostic Test: Plasma Inflammation Markers — The following blood test parameters - Tumor Necrosis Factor Alpha (TNF-α), Interleukin-6 (IL-6), and C-Reactive Protein (CRP) - will be assessed during the Screening and Day 28 visits.
Diagnostic Test: Plasma Brain-Derived Neurotrophic Facto — Plasma BDNF (Brain-Derived Neurotrophic Factor) levels will be measured during the screening and Day 28 visits.
  Other Names: Plasma BDNF
Other: Mini International Neuropsychiatric Interview — The Mini International Neuropsychiatric Interview (MINI) will be administered during the screening visit to rule out any current or past major psychiatric disorders.
  Other Names: MINI
Other: Family Psychiatric History Assessment — The Family Psychiatric History Assessment (FPHA) will be administered during the screening visit to help rule out any current or past major psychiatric disorders.
  Other Names: FPHA
Other: Beck Depression Inventory — The Beck Depression Inventory (BDI) will be administered at the following visits: screening, baseline, day 7, day 28, and day 84. It will be used to assess baseline mood and to rule out depressive symptoms.
  Other Names: BDI
Other: State-Trait Anxiety Inventory — State-Trait Anxiety Inventory (STAI) will be administered at the following visits: screening, baseline, day 7, day 28, and day 84. It will be used to screen for anxiety disorders.
  Other Names: STAI
Behavioral: Profile of Mood States — The Profile of Mood States (POMS) will be administered to assess baseline mood and emotional state.
  It will be administered at the following visits: screening, baseline, administration day, day 2, day 7, day 28, and day 84.
  On the administration day and on day 2, it will be administered at the following time points: pre-administration, and 8 and 20 hours post-administration.
  Other Names: POMS
Behavioral: Subjective Units of Distress Scale — Subjective Units of Distress Scale (SUDS) will be administered to assess anxiety and stress levels.
  It will be administered at the following visits: screening, baseline, administration day, day 2, day 7, day 28, and day 84.
  On the administration day and on day 2, it will be administered at the following time points: pre-administration, and 8 and 20 hours post-administration.
  Other Names: SUDS
Other: Five-Dimensional Altered States of Consciousness questionnaire — The Five-Dimensional Altered States of Consciousness questionnaire (5D-ASC) will be used to assess the acute subjective psychedelic experience. It will be administered after the acute effects have subsided - at 6.0 hours post-administration on the administration day, and again on day 2 - to evaluate five key experiential dimensions: visual restructuralization, oceanic boundlessness, reduction of vigilance, anxious ego dissolution, and auditory alterations. Each item will be rated using a Visual Analogue Scale (VAS) ranging from "NO, not more than usually" (0 mm) to "YES, much more than usually" (100 mm).
  Other Names: 5D-ASC
Behavioral: Integration — The integration process is conducted to support participants in processing and incorporating their therapeutic experience into daily life, with the aim of enhancing emotional insight and psychological well-being. Integration will take place at the following visits: 8.0 hours post-treatment on the administration day, day 2, day 7, day 28, and day 84.

SUMMARY:
The goal of this open-label, dose-escalation, prospective study is to evaluate the safety and psychological effects of a Psilocybin and D-Serine formulation in healthy volunteers.

The main objectives are:

1. To assess the psychological and physiological effects of psilocybin administered with D-Serine in healthy adults.
2. To determine whether D-Serine modulates or attenuates the psychedelic effects of psilocybin.
3. To evaluate the safety and tolerability of psilocybin and D-Serine co-administration.

Study population includes: 10 healthy male or female volunteers aged 25-60 years with no history of psychiatric or major medical disorders and no current evidence of such disorders.

The study includes two cohorts. The first cohort of 5 participants will receive 15 mg of Psilocybin and 5 g of D-Serine. Safety data will be collected and submitted in an interim report to the Ethics Committee. If no safety concerns arise, the second cohort will receive an increased dose of 25 mg of Psilocybin and 7 g of D-Serine to help determine the optimal dose for a future Phase IIa clinical trial.

DETAILED DESCRIPTION:
This is a first-in-human, Phase I, exploratory clinical trial designed to evaluate the safety, tolerability, and initial psychological and physiological responses to a single administration of psilocybin in combination with D-Serine in healthy adult volunteers. The rationale for this combination stems from preclinical evidence indicating that D-Serine, a naturally occurring co-agonist at the NMDA receptor, may attenuate the acute psychedelic effects of psilocybin while preserving its neuroplastic and therapeutic properties.

Preclinical studies demonstrated that D-Serine reduced the psilocybin-induced head-twitch response (HTR) in rodent models and enhanced the expression of synaptic plasticity markers (e.g., GAP43, PSD95, SV2A, synaptophysin) across multiple brain regions, with effects sustained up to 12 days post-treatment. These findings suggest that the combination may improve the safety and tolerability of psilocybin, particularly for populations sensitive to its psychoactive effects.

The trial will consist of four sequential components:

Screening Phase - to assess eligibility.

Preparation Phase - to establish therapeutic rapport and baseline assessments.

Administration Phase - involving a single oral administration of the investigational combination (psilocybin + D-Serine).

Follow-up Phase - including in-person follow-up visits on Day 2, Day 7, Day 28, and Day 84 post-treatment to monitor safety outcomes, subjective responses, and potential delayed effects.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 25-60 years, male or female.
2. Medically healthy, as confirmed by a comprehensive clinical assessment.
3. Written informed consent provided.

Exclusion Criteria:

1. History of any Axis 1 psychiatric disorder requiring pharmacotherapy such as schizophrenia, schizoaffective disorder, any other psychotic disorder, bipolar disorder, as well as non-psychotic disorders such as generalized anxiety disorder, major depressive disorder, obsessive-compulsive disorder, posttraumatic stress disorder.
2. Family history (among first-degree relatives) of schizophrenia, bipolar disorder, or other psychotic disorder
3. History of cardiovascular disorders.
4. Pregnant or breastfeeding women or women of childbearing age not using effective contraception.
5. Use of psilocybin or other psychedelic compound in the 12 months preceding the study
6. Use of medications that interact with psilocybin or D-Serine.
7. Positive urinary drug screening.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) following administration of psilocybin and D-serine | From time of dosing (Day 1) through Day 84 (final follow-up visit)
  The number, type, severity, timing, and relatedness of treatment-emergent adverse events following administration of psilocybin and D-serine. Adverse events will be assessed through continuous clinical monitoring, spontaneous reports, and structured instruments including the UKU Side Effect Rating Scale. Safety will also be evaluated via changes in vital signs, ECG, and laboratory tests (SMAC-20, CBC, urinalysis). Events will be classified using standard regulatory definitions and graded for severity and relatedness to study treatment.

SECONDARY OUTCOMES:
Change in subjective psychedelic experience measured by the 5D-ASC scale | 6 hours post-dosing and Day 2 follow-up
  Assessment of subjective altered states of consciousness using the 5-Dimensional Altered States of Consciousness scale.
  Full questionnaire consists of 94 items, each item reflects a subjective experience during the altered state.
  Each rated on a visual analog scale from 0 to 100, where:
  0 = "not at all" 100 = "extremely"
  The items are grouped into 5 empirically derived dimensions, each representing a core aspect of altered consciousness:
  Oceanic Boundlessness- Positively experienced ego dissolution, unity, bliss High scores = mystical-type experiences Anxious Ego Dissolution- Anxiety, loss of ego control, cognitive impairment High scores = difficult or fearful experiences Visionary Restructuralization -Visual imagery, hallucinations, synesthesia High scores = complex visual phenomena Auditory Alterations - Changes in auditory perception, e.g., hearing sounds or voices Reduction of Vigilance- Reduced alertness or drowsiness (less relevant in classic psychedelic states)
Change in mood states assessed by the Profile of Mood States (POMS) | Baseline, 8 and 20 hours post-dosing, Day 2, Week 1, and Day 84
  Change in emotional and mood states as measured by the POMS scale. Participants complete the questionnaire at multiple time points to evaluate transient mood fluctuations in response to treatment.
  The administered version of the POMS questionnaire consists of 28 adjectives describing various feelings and emotions, and participants rate the extent to which they have experienced each over a specified period (e.g., the past week), typically using a 5-point Likert scale ranging from 0 ("not at all") to 4 ("extremely").
Change in anxiety and stress measured by the Subjective Units of Distress Scale (SUDS) | Baseline, 8 and 20 hours post-dosing, Day 2
  Subjective assessment of distress and anxiety using the SUDS, a self-report scale ranging from 0 (no distress) to 100 (extreme distress). Assessed multiple times to track acute and residual anxiety responses.
Change in plasma D-serine concentration | Baseline and Week 1 (Day 7)
  Measurement of plasma D-serine (in micromoles per liter (µmol/L)) to explore potential neurobiological correlates of treatment. Blood collected at baseline and follow-up.
Change in plasma inflammatory markers concentration. | Baseline and Week 1 (Day 7)
  Measurement of plasma inflammatory markers to explore potential neurobiological correlates of treatment. Blood collected at baseline and follow-up.
Change in plasma BDNF concentration | Baseline and Week 1 (Day 7)
  Measurement of plasma PLASMA Brain-Derived Neurotrophic Factor (in micromoles per picograms per milliliter (pg/mL)) to explore potential neurobiological correlates of treatment. Blood collected at baseline and follow-up.
Change in plasma glutamate concentration | Baseline and Week 1 (Day 7)
  Measurement of plasma glutamate (in micromoles per liter (µmol/L)) to explore potential neurobiological correlates of treatment. Blood collected at baseline and follow-up.
Beck Depression Inventory-II (BDI-II) total score | Baseline (Day -1), Day 2, Day 7, and Day 84
  Self-reported symptoms of depression will be assessed using the 21-item Beck Depression Inventory-II, which provides a standardized index of depressive severity.
  Each corresponding to a symptom of depression, rated on a scale from 0 to 3 based on intensity. The total score ranges from 0 to 63, with higher scores indicating more severe depressive symptoms. Score interpretation is as follows: 0-13 = minimal depression, 14-19 = mild depression, 20-28 = moderate depression, and 29-63 = severe depression.
State-Trait Anxiety Inventory (STAI) - State and Trait scores | Baseline (Day -1), Day 2, Day 7, and Day 84
  Anxiety symptoms will be measured using the STAI, which provides separate scores for State Anxiety (how participants feel in the moment) and Trait Anxiety (how they generally feel).
  The STAI consists of 40 items - 20 assessing state anxiety and 20 assessing trait anxiety - each rated on a 4-point Likert scale. Scores for each subscale range from 20 to 80, with higher scores indicating greater levels of anxiety. Generally, a score of 20-37 suggests low anxiety, 38-44 moderate anxiety, and 45-80 high anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel